CLINICAL TRIAL: NCT02456103
Title: Phase 3 Extension Study of Ataluren (PTC124) in Patients With Nonsense Mutation Cystic Fibrosis
Brief Title: Extension Study of Ataluren in Participants With Nonsense Mutation Cystic Fibrosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Cystic Fibrosis (CF) data from the double-blind CF Study PTC124-GD-021-CF did not meet endpoints.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-021e-CF
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ataluren (Experimental): Participants will be administered ataluren orally at a dose of 10 milligrams/grams (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for up to 96 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with water or milk.
  Other Names: PTC124; Translarna

SUMMARY:
This is an open-label extension study for participants who completed a Phase 3, placebo-controlled study of ataluren in participants with nonsense mutation cystic fibrosis (nmCF) not receiving chronic inhaled aminoglycosides.

DETAILED DESCRIPTION:
The primary objective of this Phase 3 extension study will be to obtain long-term safety data to augment the overall safety database. The secondary objectives will be to augment the efficacy data collected in the double-blind study (PTC124-GD-021-CF; NCT02139306).

ELIGIBILITY:
Inclusion Criteria:

* Completion of study treatment (placebo or active) in the previous Phase 3, double-blind study protocol (Protocol PTC124-GD-021-CF)
* Evidence of signed and dated informed consent/assent document(s) indicating that the participant (and/or the participant's parent/legal guardian) has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug.
* Ongoing participation in any other therapeutic clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McIntosh, MD, Study Director — PTC Therapeutics
Locations (70):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Stanford University-Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center, Tyler, Texas
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Argentina (2):
  - Hospital de Ninos Ricardo Gutierrez, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Chermside
  - Princess Margaret Hospital, Perth
- Belgium (3):
  - University Hospital Brussels, Brussels
  - Hopital Universitaire des Enfants Reine Fabiola, Brussels
  - University Hospital Leuven, Leuven
- Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul, Porto Alegre, Brazil
- Bulgaria (2):
  - University Mulitiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
- Canada (3):
  - Clinical Research Institute of Montreal, Montreal
  - University of Toronto Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- France (4):
  - Hoptial Arnaud de Villeneuve, Montpellier
  - Hopital Necker - Enfants Malades, Paris
  - Centre de Perharidy, Roscoff
  - Centre Hospitalier Regional Sud Reunion, Saint-Pierre
- Germany (7):
  - Charite-Universitatsmedizin Berlin, Berlin
  - St. Josef Hospital GmbH, Bochum
  - University of Cologne Children's Hospital, Cologne
  - Christiane Herzog CF-Zentrum, Frankfurt am Main
  - Universitatsklinikum Jena, Jena
  - LMU Klinikum der Universitat Muchen, Munich
  - Dr. Von Haunersches Kinderspital, München
- Ippokratio General Hospital Of Thessaloniki, Thessaloniki, Greece
- Israel (2):
  - Meyer Children's Hospital, Haifa
  - Hadassah University Hospital, Jerusalem
- Italy (6):
  - Azienda Ospedaliero Universitaria Ospedall Riuniti di Acona-Umberto I G.M. Lancisi G. Salesi, Ancona
  - Azienda Ospedaliera A Meyer, Florence
  - Lombardia Cystic Fibrosis Center, Milan
  - Azienda Policlinico Umberto I, Rome
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Azienda Ospedaliera di Verona, Verona
- Netherlands (2):
  - Hagaziekenhuis, s-Gravenweg, South Holland
  - Radboud University, Nijmegen
- Poland (2):
  - Szpital Dzieciecy Polanki im Macieja Plazynskiego w Gdansku, Gdansk
  - Institute of Mother and Child, Warsaw
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital University, Barcelona
  - Hospital San Juan, Esplugues de Llobregat
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital de Sabadell, Consorci Sanitari Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - St James University Hospital, Leeds
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible participants, including those who received placebo in the double-blind study (PTC124-GD-021-CF; NCT02139306), were enrolled to this open-label extension study. To avoid interruption in treatment, when possible, Screening/Baseline for this extension study was to occur on the same day as the End-of-Study visit for the double-blind study.
Groups:
- Ataluren: Participants were administered ataluren orally at a dose of 10 milligrams/grams (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for up to 96 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 246
As-Treated Population (Participants who received at least 1 dose of ataluren.) | 245
Intent-to-treat (ITT) Population (Participants in the As-Treated Population with at least 1 postbaseline efficacy assessment.) | 244
Completed | 0
Not Completed | 246
Not completed — Study Closure | 207
Not completed — Physician Decision | 1
Not completed — Required prohibited medications | 5
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 5
Not completed — Abnormal Laboratory Value | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 24

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of ataluren (As-Treated Population).
Groups:
- Ataluren: Participants were administered ataluren orally at a dose of 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for up to 96 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 132
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4
  White | 235
  White-Arabic/North African Heritage | 1
  Non-White | 5
  Hispanic or Latino | 16
  Not Hispanic or Latino | 229

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAE: any untoward medical occurrence or undesirable event that begins or worsens following administration of study drug, whether or not considered related to study drug by Investigator. Serious adverse event (SAE): an adverse event (AE) resulting in any of following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying) or persistent or significant disability/incapacity. Except for cystic fibrosis (CF) pulmonary exacerbations, an event wasn't reported as an SAE, if event was exclusively a relapse or an expected change or progression of baseline CF. AEs included both SAEs and nonserious AEs. AEs classified according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 and coded using Medical Dictionary for Regulatory Activities. A summary of SAEs and all nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to Week 100
Population: Participants who received at least 1 dose of ataluren (As-Treated Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 245
Participants
  At least 1 TEAE | 222
  Mild TEAE | 28
  Moderate TEAE | 147
  Severe TEAE | 46
  Life-Threatening TEAE | 1
  Fatal TEAE | 0
  Serious TEAE | 89
  TEAE Unrelated to Study Drug | 140
  TEAE Unlikely Related to Study Drug | 55
  TEAE Possibly Related to Study Drug | 23
  TEAE Probably Related to Study Drug | 4

2. Primary Outcome: Number of Participants With a Clinically Meaningful Abnormal Clinical Laboratory (Serum Biochemistry, Hematology, and Urinalysis) Parameter
Description: Clinical laboratory results considered clinically meaningful were determined by Investigator. Serum biochemistry parameters: sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, magnesium, calcium, phosphorus, uric acid, glucose, total protein, albumin, globulin, bilirubin, creatine kinase, lactate dehydrogenase, alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, alkaline phosphatase, total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides, and cystatin C. Hematology parameters: white blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, red cell count with morphology, and platelet count. Urinalysis parameters: pH, specific gravity, glucose, ketones, blood, protein, creatinine, urobilinogen, bilirubin, nitrite, and leukocyte esterase. A summary of all SAEs/nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to Week 100
Population: Participants who received at least 1 dose of ataluren (As-Treated Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 245
Participants | 0

3. Secondary Outcome: Change From Baseline in Percent-Predicted Forced Expiratory Volume in 1 Second (FEV1) as Measured by Spirometry at Week 24
Description: Pulmonary function of percent-predicted FEV1 was measured using a spirometer. FEV1 is the volume of air that can forcibly be blown out in 1 second. Each percent-predicted FEV1 was based gender, age, and the height value obtained at the same study visit. The percentage of change in percent-predicted of FEV1 was calculated as follows: (percent-predicted FEV1 - Baseline percent-predicted FEV1/Baseline percent-predicted FEV1)*100.
Time Frame: Baseline, Week 24
Population: Participants who received at least 1 dose of ataluren and have at least 1 postbaseline efficacy assessment (ITT Population) and had evaluable FEV1 data.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Ataluren
Number analyzed (Participants) | 233
percentage of predicted FEV1
  Baseline | 60.219 (17.6163)
  Change from Baseline at Week 24: number analyzed (Participants) | 205
  Change from Baseline at Week 24 | 0.015 (6.7180)

4. Secondary Outcome: Change From Baseline in Percent-Predicted of Forced Vital Capacity (FVC) as Measured by Spirometry at Week 24
Description: Pulmonary function of FVC was measured using a spirometer. FVC is the volume of air that can forcibly be blown out. Each percent-predicted FVC was based gender, age, and the height value obtained at the same study visit. The percentage of change in percent-predicted of FVC was calculated as follows: (percent-predicted FVC - Baseline percent-predicted FVC/Baseline percent-predicted FVC)*100.
Time Frame: Baseline, Week 24
Population: Participants who received at least 1 dose of ataluren and have at least 1 postbaseline efficacy assessment (ITT Population) and had evaluable FVC data.
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Ataluren
Number analyzed (Participants) | 233
percentage of predicted FVC
  Baseline | 75.249 (15.8508)
  Change from Baseline at Week 24: number analyzed (Participants) | 205
  Change from Baseline at Week 24 | 0.166 (6.5276)

5. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Between 25% and 75% of Expiration (FEF25-75) as Measured by Spirometry at Week 24
Description: Pulmonary function of FEF25-75 was measured using a spirometer. FEF25-75 is the forced expiratory flow between 25% and 75% of vital capacity. Each percent-predicted FEF25-75 was based gender, age, and the height value obtained at the same study visit. The percentage of change in percent-predicted of FEF25-75 was calculated as follows: (percent-predicted FEF25-75 - Baseline percent-predicted FEF25-75/Baseline percent-predicted FEF25-75)*100.
Time Frame: Baseline, Week 24
Population: Participants who received at least 1 dose of ataluren and have at least 1 postbaseline efficacy assessment (ITT Population) and had evaluable FEF25-75 data.
Measure: Mean (Standard Deviation); unit: percentage of FEF25-75
Arm/Group | Ataluren
Number analyzed (Participants) | 233
percentage of FEF25-75
  Baseline | 38.099 (22.0980)
  Change from Baseline at Week 24: number analyzed (Participants) | 205
  Change from Baseline at Week 24 | 0.698 (13.1241)

6. Secondary Outcome: Rate of Pulmonary Exacerbations as Defined by Modified Fuch's Criteria Over 48 Weeks
Description: A modified Fuchs' exacerbation was defined as an event requiring treatment with or without intravenous antibiotics for any 4 of the following 12 symptoms: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10 percent or more from a previously recorded value; or radiographic changes indicative of pulmonary function. The 48-week rate = (the total number of events/ treatment duration by week)*48.
Time Frame: Baseline up to Week 48
Population: Participants who received at least 1 dose of ataluren and have at least 1 postbaseline efficacy assessment (ITT Population).
Measure: Mean (Standard Deviation); unit: exacerbations
Arm/Group | Ataluren
Number analyzed (Participants) | 244
exacerbations | 1.051 (2.1654)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 100
Description: Adverse events collected from participants who received at least 1 dose of ataluren (As-Treated Population).
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 1/245
Serious Adverse Events (participants affected / at risk) | 89/245
Other Adverse Events (participants affected / at risk) | 191/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ataluren (N=245)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 63
Mycobacterium abscessus infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral pericarditis (Infections and infestations) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Forced expiratory volume decreased (Investigations) | 2
Protein urine present (Investigations) | 1
Pseudomonas test positive (Investigations) | 1
Pulmonary function test decreased (Investigations) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/113 — This is a sex-specific adverse event that only affects female participants.
Depressed level of consciousness (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/113 — This is a sex-specific adverse event that only affects female participants.
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=245)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 136
Influenza (Infections and infestations) | 13
Sinusitis (Infections and infestations) | 25
Upper respiratory tract infection (Infections and infestations) | 21
Viral upper respiratory tract infection (Infections and infestations) | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 32
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 14
Forced expiratory volume decreased (Investigations) | 16
Headache (Nervous system disorders) | 16
Nausea (Gastrointestinal disorders) | 14
Pyrexia (General disorders) | 13

LIMITATIONS AND CAVEATS:
This study was terminated early because the CF data from the double-blind CF Study PTC124-GD-021-CF (NCT02139306) did not meet endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the Sponsor for review. The Sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-03-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT02456103/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT02456103/SAP_001.pdf